CLINICAL TRIAL: NCT05325957
Title: Effects of Norepinephrine and Volume Expansion in Capillary Refill Time in Septic Shock in Angers University Hospital
Acronym: NOVECAR-A
Status: Withdrawn | Type: Observational
Why Stopped: Canadian study completed before beginning of French study sites
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC22_0096
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Norepinephrine variation: Patients with septic shock, cardiac output monitoring device with the PICCO2 system or swan ganz catheter and decision by the physician in charge to modify the norepinephrine dose.
- Fluid infusion: Patients with septic shock, cardiac output monitoring device with the PICCO2 system or swan ganz catheter and decision by the physician in charge to give fluid infusion

SUMMARY:
the purpose of this study is to assess the effect of norepinephrine and fluid expansion on capillary refill time during septic shock.

DETAILED DESCRIPTION:
An interventional study compared, in septic shock, the effect of resuscitation strategy targeting normalization of capillary refill time versus strategy targeting serum lactate level. This last highlight a decrease of organ dysfunction at 72 hours with capillary refill time strategy and non-significant trend towards lower 28-day mortality in the capillary refill time strategy group.

The strategy guided by the decreasing of capillary refill time allowed the administration of less fluid than that guided by lactate. This is an important advantage when the intensive care doctor know that the mortality of patient in septic shock increases with the amount of fluid administered.

However, the variations of capillary refill time induced by the principal treatment in septic shock (norepinephrine and fluid resuscitation) during circulatory failure are actually insufficiently described. The purpose of this study is to assess the effect of norepinephrine and fluid expansion on capillary refill time during septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock
* Presence of a cardiac output monitoring
* Decision by the physician in charge to perform vascular filling or modification the norepinephrine dose

Exclusion Criteria:

* Patient under a tutelage measure or placed under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock, cardiac output monitoring device with the PICCO2 system or swan ganz catheter
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Difference of capillary refill time before and after the therapeutic change | Change from capillary refill time between the 15 min before the therapeutic, Immediately after fluid administration and within the 15 minutes of a change in norepinephrine dose
  Capillary refill time (CRT) is time required for return of color after application of blanching pressure to a distal capillary bed. In this study, we made a calibrated compression of the skin using a piston for seven seconds, and we recorded CRT with a smartphone's video camera.

SECONDARY OUTCOMES:
Correlation between capillary refill time and perfusion index | Change from capillary refill time between the 15 min before the therapeutic, Immediately after fluid administration and within the 15 minutes of a change in norepinephrine dose
  Capillary refill time is time required for return of color after application of blanching pressure to a distal capillary bed. In this study, we made a calibrated compression of the skin using a piston for seven seconds, and we recorded CRT with a smartphone's video camera.
Least significant change of capillary refill time | Change from capillary refill time between the 15 min before the therapeutic, Immediately after fluid administration and within the 15 minutes of a change in norepinephrine dose
  Capillary refill time is time required for return of color after application of blanching pressure to a distal capillary bed. In this study, we made a calibrated compression of the skin using a piston for seven seconds, and we recorded CRT with a smartphone's video camera.
Difference between capillary refill time on thorax and on the index finger tip | Change from capillary refill time between the 15 min before the therapeutic, Immediately after fluid administration and within the 15 minutes of a change in norepinephrine dose
  Capillary refill time is time required for return of color after application of blanching pressure to a distal capillary bed. In this study, we made a calibrated compression of the skin using a piston for seven seconds, and we recorded CRT with a smartphone's video camera

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ASFAR, M.D- Ph.D, Principal Investigator — Angers CHU
Locations (1):
- Medical Intensive Care Unit, Angers, Maine-et-Loire, France

IPD SHARING:
Plan to Share IPD: Undecided